CLINICAL TRIAL: NCT07024888
Title: Effect of Food on the Pharmacokinetics of SSS17 Capsules: A Study in Chinese Healthy Subjects
Brief Title: A Study Evaluating the Food Effect on the Pharmacokinetics of SSS17 Capsules in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: SSS17-103
Record Dates: First submitted 2025-06-05; First posted 2025-06-17 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Healthy Subjects (HS)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fasting Group (Other)
  Interventions: Drug: SSS17
- Low-fat Meal Concomitant Administration Group (Other)
  Interventions: Drug: SSS17
- High-fat Meal 2-Hour Post-dose Group (Other)
  Interventions: Drug: SSS17

INTERVENTIONS:
Drug: SSS17 — Single oral administration of SSS17

SUMMARY:
This study mainly compared the blood drug concentration and main pharmacokinetic parameters of SSS17 capsules taken orally once by healthy Chinese subjects under fasting conditions, 2 hours after administration, and when consuming a high-fat meal or a low-fat meal simultaneously. The study evaluated the impact of food on SSS17 capsules.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subjects aged 18 to 45 years
2. Good health status with no clinically significant medical history.
3. Agreement to use effective contraception from signing ICF until 6 months after trial completion, with no reproductive plan.
4. Voluntarily sign informed consent form (ICF), capable of protocol compliance and scheduled follow-up

Exclusion Criteria:

1. Hypersensitivity to investigational drug/excipients.
2. Dysphagia, GI disorders affecting absorption, or relevant surgery history .
3. Intolerance to venipuncture or needle/blood phobia.
4. Clinically significant disorders affecting drug ADME.
5. Clinically significant abnormalities in vital signs/PE/labs/12-lead ECG/chest X-ray at screening.
6. Family history of malignancy or major surgery within 3 months pre-screening.
7. Participation in other drug/device trials with investigational product use within 3 months.
8. Blood donation/loss within 3 months.
9. Special diets (pitaya/grapefruit products) or strenuous exercise within 7 days pre-dosing affecting ADME.
10. Any medication use within 14 days pre-dosing.
11. Regular alcohol >14 units/week within 3 months.
12. Smoking >5 cigarettes/day within 3 months or unwilling to abstain during trial.
13. Caffeine products within 48h pre-dosing.
14. Alcohol consumption within 48h or positive alcohol screen.
15. Positive serology for HBsAg, HCV Ab, HIV Ab, or syphilis.
16. Pregnancy/lactation or unprotected sex
17. Positive drug screen, drug abuse history, or drug use within 3 months.
18. Any condition compromising safety/compliance, or investigator's judgment of unsuitability

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-03-16 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Cmax | Day1 to Day73
AUC | Day 1 to Day 73

SECONDARY OUTCOMES:
Tmax | Day1 to Day73
t1/2 | Day 1 to Day 73
CL/F | Day 1 to Day 73
AEs | up to Day 73

CONTACTS AND LOCATIONS:
Locations (1):
- The Affilated Hospital Of QingDao University, Qingdao, China

IPD SHARING:
Plan to Share IPD: Undecided